CLINICAL TRIAL: NCT03080961
Title: The VIBLOK SAfety and perFormancE Trial
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CLJI Worldwide (Industry)
Collaborators: Applied Clinical Services BV (Unknown); UMC Utrecht (Other); University of Rotterdam, The Netherlands (Other); University of Washington (Other); EB FlevoResearch BV (Unknown); PreCare Trial & Recruitment B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-01
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-10

CONDITIONS: HSV-2 Infection; Genital Herpes
Keywords: Barrier cream
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Intervention Model Description: Trial participants take extra-genital swabs before and after application of the barrier cream.
Masking Description: Vials with the sample will be coded. The assessor does not know the coding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before and after VIBLOK (Experimental): The degree to which HSV-2 is blocked by the VIBLOK cream is determined by comparing the amount of HSV in the external genital area before and after application of the cream. So participants are their own control.
  Interventions: Device: VIBLOK barrier cream

INTERVENTIONS:
Device: VIBLOK barrier cream — VIBLOK safety and performance has not been proven yet in humans with an HSV-2 infection.

SUMMARY:
Genital herpes has a high prevalence in industrialized as well as developing countries.

Genital herpes causes genital ulcers, increases risk for acquiring HIV infection, and may be transmitted mother to child during birth with possible serious consequences.

Medical treatments and condoms only partially reduce the risk for transmission from/ to sexual partners. Genital herpes transmission despite use of condoms is thought to be due to transfer via skin-to-skin contact in unprotected areas, and HSV-2 transmission may be enhanced by current shaving habits in the genital area leading to micro lesions (lacerations) of the skin.

VIBLOK™ is a cream designed to impede the passage of viruses, such as HSV-2, across the skin. Bench and animal experiments indicate that it can block virus transmission such as HSV-2 over 80%.

The objective of the SAFE trial is to assess the safety and performance of VIBLOK in adults with HSV-2 infection by comparing virus detection in the extra-genital area before and after application of the barrier cream.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female and at least 18 years of age
2. HSV-2 seropositive by the UW Western blot or Alegria assay
3. History of recurrent genital herpes with at least 3 recurrences in the last year or, if currently on suppressive/ prophylactic therapy, prior to starting the therapy (antiviral therapy has to be stopped at least 7 days prior to initiation of the trial product).
4. General good health at the discretion of the investigator.
5. Willing to not use any topical genital therapy aside from the study device for the duration of the trial.
6. Willing to not use any systemic anti HSV therapy during the entire study starting 7 days prior to baseline.
7. Willing to obtain 2 swabs from external-genital areas once daily for the duration of the trial.
8. Willing to keep a daily trial diary during the treatment period.
9. Negative pregnancy test for women at screening.
10. Willing to use contraceptives for the duration of the study.
11. Subject must be willing and able (in the opinion of the investigator) to understand the patient information and informed consent form and to comply with the clinical trial protocol and procedures.
12. Subject must be willing to give written informed consent.

Exclusion Criteria:

1. Serious medical conditions, such as diabetes, significant autoimmune disease, cancer or immunosuppression, etc. that at the discretion of the investigator will likely affect study outcomes
2. Treatment with systemic steroids or other immune-modulating agents
3. Participation in any investigational drug or device trial within 30 days prior to screening.
4. Pregnancy or breastfeeding, in case of women.
5. Any other conditions that in the judgment of the investigator would preclude successful completion of the clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivienne vd Walle, MD, Principal Investigator — PreCare Trial & Recruitment B.V.
Locations (3):
- Netherlands (3):
  - EB FlevoResearch, Almere Stad, Flevoland
  - PT&R, Beek, Limburg
  - EB UtrechtResearch, Utrecht

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon written informed consent, 82 subjects were enrolled based on their medical history of recurrent genital herpes.
Pre-assignment Details: Of the 82 subjects enrolled, 46 had a confirmed HSV-2 infection and started applying VIBLOK.
Groups:
- Treatment Group: 46 subjects with a confirmed HSV-2 infection, took external genital skin swabs before and after applying minimally 0.8 pack (~4 ml) of VIBLOK per swab session.
Period: Overall Study
Arm/Group | Treatment Group
Started | 46
Completed | 43
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Adults with recurrent genital herpes due to an HSV-2 infection and that applied VIBLOK at least once.
Groups:
- As Treated Population: Participants that applied VIBLOK at least once
Arm/Group | As Treated Population
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 2
  Unknown or Not Reported | 7
HSV-1 co-infection [Count of Participants; unit: Participants] | 15
Number of recurrences past year [Mean (Standard Deviation); unit: episodes] | 5.7 (2.60)
Years since diagnosis genital herpes [Mean (Standard Deviation); unit: years] | 5.8 (6.26)

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Device Effects
Description: Percentage SADE's in the as treated population.
Time Frame: 26-32 days
Population: 46 eligible subjects that applied VIBLOK for an average of 27.2 days.
Measure: Number (95% Confidence Interval); unit: Percentage SADE's
Groups:
- During VIBLOK Application: Percentage SADE's in subjects applying VIBLOK for a minimum of 26 days.
Arm/Group | During VIBLOK Application
Number analyzed (Participants) | 46
Percentage SADE's | 0 [0 to 7.7]
Statistical Analysis 1: Comparison: During VIBLOK Application; SADE rate after minimally 26 days of VIBLOK treatment will be assessed by calculating the upper limit of the 2-sided exact 95% Clopper-Pearson confidence interval which needs to be below 10%. With a sample size of 36, an exact two-sided 95.0% confidence interval for a single proportion would show that the SADE incidence is below 10% at an expected incidence of 0.1%; Test type: Other; SADE percentage = 0, 95% CI 2-sided [0.0 to 7.7]

2. Secondary Outcome: HSV-2 Detection Rate in AT Population
Description: Change in HSV-2 detection rate on days with asymptomatic shedding after applying VIBLOK.
Time Frame: 26-32 days
Population: 45 subjects that returned swabs before and after VIBLOK application.
Measure: Mean (95% Confidence Interval); unit: Mean number of swabs with shedding
Groups:
- Before VIBLOK: Days with HSV detection in the external genital area before application of VIBLOK.
- After VIBLOK: Days with HSV detection in the external genital area after application of VIBLOK.
Arm/Group | Before VIBLOK | After VIBLOK
Number analyzed (Participants) | 45 | 45
Mean number of swabs with shedding | 2.9 [1.7 to 4.1] | 2.6 [1.4 to 3.8]
Statistical Analysis 1: Comparison: Before VIBLOK vs After VIBLOK; Statistical analysis will evaluate the difference in detection rate between pre and post-VIBLOK swabs. For each person the number of swabs with shedding only pre-VIBLOK will be assessed, and then the number of swabs with shedding only post-VIBLOK will be subtracted. A number above 0 indicates a decreased detection rate after VIBLOK. With an 8% anticipated asymptomatic shedding rate, 80% power, 50 subjects taking samples for 28 days are needed to show a 50% reduction; Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: HSV-2 Copy Number in AT Population
Description: Change in HSV-2 copy number on days with asymptomatic shedding after applying VIBLOK.
Time Frame: 26-32 days
Population: A total of 25 out of 46 subjects in the AT population had days with asymptomatic HSV shedding.
Measure: Mean (95% Confidence Interval); unit: HSV copy number
Groups:
- Before VIBLOK: HSV amount in external genital swabs on days with asymptomatic shedding before applying VIBLOK.
- After VIBLOK: HSV amount in external genital swabs on days with asymptomatic shedding after applying VIBLOK.
Arm/Group | Before VIBLOK | After VIBLOK
Number analyzed (Participants) | 25 | 25
HSV copy number | 100446.2 [24623.8 to 176268.7] | 43691.8 [1954.4 to 85429.2]
Statistical Analysis 1: Comparison: Before VIBLOK vs After VIBLOK; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: ADE Description
Description: Nature and frequency of (possible) device related adverse events.
Time Frame: 1-33 days
Population: AT Population that applied VIBLOK at least once.
Measure: Number; unit: Count of participants per ADE type
Groups:
- During VIBLOK Application: Subjects that applied VIBLOK at least once.
Arm/Group | During VIBLOK Application
Number analyzed (Participants) | 46
Count of participants per ADE type
  Toxic reaction | 0
  Possible allergic reaction | 2
  Itching/tingling/burning sensation | 19
  Infection | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first day of VIBLOK application until 30 days after the last visit to the research clinic.
Description: Definitions are applied conform ISO 14155; 2011.
Groups:
- During VIBLOK Application: All AEs were recorded in subjects in all subjects applying VIBLOK at least once until 30 days after the last visit to the research clinic.
Arm/Group | During VIBLOK Application
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 39/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | During VIBLOK Application (N=46)
Toxic reaction (Injury, poisoning and procedural complications) | 0 (0)
Possible device related allergic reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Itching/tingling/burning sensation (Skin and subcutaneous tissue disorders) | 19 (21)
HSV recurrence (Skin and subcutaneous tissue disorders) | 19 (29)
Not-device related infection (Infections and infestations) | 11 (16)
Possible not-device related allergic reaction (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Other, undefined (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03080961/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03080961/SAP_001.pdf